CLINICAL TRIAL: NCT04409873
Title: Effect of Antiseptic Mouthwash/Gargling Solutions and Pre-procedural Rinse on SARS-CoV-2 Load (COVID-19)
Brief Title: Antiseptic Mouthwash / Pre-Procedural Rinse on SARS-CoV-2 Load (COVID-19)
Acronym: AMPoL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The funder decided not to continue funding, causing enrollment to cease prematurely and curtailing originally planned analyses. Participants with any samples collected after the baseline pre-rinse samples were included in the analysis.
Sponsor: University of California, San Francisco (Other)
Collaborators: Rowpar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20-30874; R00RG2901 (Other Grant/Funding Number: UCOP Emergency COVID19 Rsrch Fd: Cal Breast Cancer Rsrch Pgm)
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: COVID-19; SARS-CoV 2; Severe Acute Respiratory Syndrome Coronavirus 2; Virus Disease; Coronavirus Infections; Pharyngeal Diseases
Keywords: Anti-Infective Agents, Local; Mouthwashes; Gargle; Saliva
MeSH Terms: conditions — COVID-19; Virus Diseases; Coronavirus Infections; Pharyngeal Diseases | interventions — Hydrogen Peroxide; Cetylpyridinium; chlorine dioxide; Water; Ethanol

STUDY DESIGN:
Intervention Model Description: A blinded randomized controlled parallel group design trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Study participants will be blinded to the solutions to the extent possible (i.e., similar packages with identification number bar codes).
  The lab technician who evaluates the SARS-CoV-2 load in samples will be blinded to the solutions and study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Control (Distilled Water) (Placebo Comparator): Over the counter: Distilled water
  Interventions: Drug: Distilled water
- Oral-B Mouth Sore (H2O2) mouthwash (Experimental): Over the counter: Oral-B Mouth Sore (Oral-B, USA) contains hydrogen peroxide (H2O2)
  Interventions: Drug: Oral-B Mouth Sore mouthwash
- Crest Pro-Health Multi-Protection (C21H38ClN) mouthwash (Experimental): Over the counter: Crest Pro-Health Multi-Protection (Crest, USA) contains cetylpyridinium chloride (C21H38ClN)
  Interventions: Drug: Crest Pro-Health Multi-Protection mouthwash
- CloSYS (ClO2) mouthwash (Experimental): Over the counter: CloSYS Ultra Sensitive Rinse (Rowpar Pharmaceutical Inc., USA) contains stabilized chlorine dioxide (ClO2)
  Interventions: Drug: CloSYS Ultra Sensitive Rinse mouthwash
- Listerine Mouthwash (Experimental): Over the counter: Listerine Zero (Alcohol-Free)(Johnson and Johnson, USA) (C30H52O3)
  Interventions: Drug: Listerine Zero Mouthwash Product

INTERVENTIONS:
Drug: Oral-B Mouth Sore mouthwash — Rinse and gargle 4 times daily, for 60 seconds, for 4 weeks.
  Other Names: hydrogen peroxide; H2O2
  Arms: Oral-B Mouth Sore (H2O2) mouthwash
Drug: Crest Pro-Health Multi-Protection mouthwash — Rinse and gargle 4 times daily, for 60 seconds, for 4 weeks.
  Other Names: cetylpyridinium chloride; C21H38ClN
  Arms: Crest Pro-Health Multi-Protection (C21H38ClN) mouthwash
Drug: CloSYS Ultra Sensitive Rinse mouthwash — Rinse and gargle 4 times daily, for 45 seconds, for 4 weeks.
  Other Names: chlorine dioxide; ClO2
  Arms: CloSYS (ClO2) mouthwash
Drug: Distilled water — Rinse and gargle 4 times daily, for 60 seconds, for 4 weeks.
  Other Names: water; H2O
  Arms: Control (Distilled Water)
Drug: Listerine Zero Mouthwash Product — Rinse and gargle 4 times daily, for 30 seconds, for 4 weeks.
  Other Names: alcohol-free
  Arms: Listerine Mouthwash

SUMMARY:
In this pilot trial, 150 confirmed COVID-19 individuals will be randomly assigned to 1 of 5 groups: distilled water, CloSYS Ultra Sensitive Rinse (Rowpar Pharmaceutical Inc., USA), Oral-B Mouth Sore (Oral-B, USA), Crest Pro-Health Multi-Protection (Crest, USA), or Listerine Zero (Johnson and Johnson, USA).

Study participants will be asked to rinse/gargle with 10-20ml (according to the rinse instructions) of the assigned solutions 4 times per day, for 30-60 seconds, for 4 weeks.

DETAILED DESCRIPTION:
SARS-CoV-2, the virus causing COVID-19, has affected vulnerable individuals, especially those with comorbidities, and high exposure health care workers (HCWs). Typically, the virus first colonizes in the upper respiratory tract (URT) causing clinical symptoms such as coughing, sore throat, and then is transferred to the lower respiratory tract (LRT) which can lead to severe pneumonia, acute respiratory distress syndrome (ARDS), sepsis, and death, if it is not managed.

The World Health Organization (WHO) has presented comprehensive guidelines underscoring personal hygiene measures including respiratory hygiene against SARS, MERS, influenza, and now SARS-CoV-2 / COVID-19. While personal protection equipment (PPE), personal hygiene measures, environmental infection control, and physical distancing are crucial in mitigating disease transmission, respiratory hygiene measures do not prevent SARS-CoV-2 colonization in URTs and LRTs of infected individuals (symptomatic and asymptomatic).

Experimental and clinical research studies on infections similar to COVID-19 such as SARS, MERS, and H5N1 have shown that using antiseptic mouthwash/gargling solutions, such as products containing chlorhexidine gluconate (CHG), polyvinylpyrrolidone iodine (PVP-I), chlorine dioxide (ClO2), cetylpyridinium chloride (CPC), and hydrogen peroxide (H2O2) can reduce viral load. A randomized controlled trial (N=387) showed efficacy and cost-effectiveness of gargling with water or a product containing PVP-I (3X/day, 20 seconds) on URTIs in healthy volunteers (18-65 years) over 60 days from a societal perspective; in vitro studies have shown that CloSYS, an over the counter mouthwash containing ClO2, was effective on inactivating SARS-CoV as well as disinfecting dental unit waterlines, and biofilm control in ultrasonic dental scaling units. A recent study has shown that CloSYS Ultra Sensitive Oral Rinse reduced the viral load of SARS CoV 2, SARS CoV, and Influenza A H3N2 to a varying extent. The data show that the viral load reduction of SARS CoV 2 by Ultra Sensitive rinse was 10 fold more than the reduction of SARS CoV in 30s. Recently, the US Centers for Disease Control (CDC) and the American Dental Association (ADA) have recommended using a mouthwash containing 1.0-1.5% H2O2 as a pre-procedural rinse before dental treatment to potentially reduce SARS-CoV-2 load; however, no in vivo clinical studies have been conducted to support this claim.

The aim of this pilot trial is to evaluate the effect of four over-the-counter antiseptic mouthwash/gargling solutions compared to a control (distilled water) to reduce SARS-CoV-2 load. In addition, study participants will be assessed for the severity of their clinical symptoms during the study period. The 4-week protocol was selected as studies have shown that patients can continue to shed the virus and potentially transmit it to the others for a 2 to 4 week period. An interim analysis is planned when 10 participants per arm (50 total) complete the study using the alpha-spending function with O'Brien-Fleming boundary rule.

ELIGIBILITY:
Inclusion Criteria:

* Tested positive for COVID-19 with a sample collected in the prior 7 days
* Ability to read and speak English or Spanish
* Ability to participate in the study for 4 weeks
* Being asymptomatic or having mild or moderate symptoms (for example, sore throat, coughing, fever, fatigue)
* Ability to rinse/gargle
* Not having any condition that might worsen with gargling solutions
* Not having a history of mouthwash sensitivity
* Not having an allergy to any mouthwash that has been used before
* Not using another mouthwash/gargling solution since the most recent positive test
* Not taking antimicrobial medications (antibacterial, antiviral, antibiotics including off-label FDA-approved medications such as hydroxychloroquine)
* Anticipated ability to participate in the study for 4 weeks
* Have a cellphone and agree to receive text messages for reminders to use mouthwash during the day and for follow-up visits, and can videoconference (like zoom) on a cellphone, tablet, or computer for sample collection instructions

Exclusion Criteria:

* People who because of their symptoms intend to receive antiviral medications that could potentially affect viral load in their saliva samples
* Pregnant or lactating women due to potential aversions to mouthwash solution taste/smell.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2022-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Gansky, DrPH, Principal Investigator — Professor and Lee Hysan Chair of Oral Epidemiology
Locations (1):
- University Of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Meng L, Hua F, Bian Z. Coronavirus Disease 2019 (COVID-19): Emerging and Future Challenges for Dental and Oral Medicine. J Dent Res. 2020 May;99(5):481-487. doi: 10.1177/0022034520914246. Epub 2020 Mar 12. PMID 32162995
- [Background] Xu J, Li Y, Gan F, Du Y, Yao Y. Salivary Glands: Potential Reservoirs for COVID-19 Asymptomatic Infection. J Dent Res. 2020 Jul;99(8):989. doi: 10.1177/0022034520918518. Epub 2020 Apr 9. No abstract available. PMID 32271653
- [Background] Reimer K, Wichelhaus TA, Schafer V, Rudolph P, Kramer A, Wutzler P, Ganzer D, Fleischer W. Antimicrobial effectiveness of povidone-iodine and consequences for new application areas. Dermatology. 2002;204 Suppl 1:114-20. doi: 10.1159/000057738. PMID 12011534
- [Background] Nagatake T, Ahmed K, Oishi K. Prevention of respiratory infections by povidone-iodine gargle. Dermatology. 2002;204 Suppl 1:32-6. doi: 10.1159/000057722. PMID 12011518
- [Background] Eggers M, Koburger-Janssen T, Eickmann M, Zorn J. In Vitro Bactericidal and Virucidal Efficacy of Povidone-Iodine Gargle/Mouthwash Against Respiratory and Oral Tract Pathogens. Infect Dis Ther. 2018 Jun;7(2):249-259. doi: 10.1007/s40121-018-0200-7. Epub 2018 Apr 9. PMID 29633177
- [Background] Sakai M, Shimbo T, Omata K, Takahashi Y, Satomura K, Kitamura T, Kawamura T, Baba H, Yoshihara M, Itoh H; Great Cold Investigators-I. Cost-effectiveness of gargling for the prevention of upper respiratory tract infections. BMC Health Serv Res. 2008 Dec 16;8:258. doi: 10.1186/1472-6963-8-258. PMID 19087312
- [Background] Wang WK, Chen SY, Liu IJ, Chen YC, Chen HL, Yang CF, Chen PJ, Yeh SH, Kao CL, Huang LM, Hsueh PR, Wang JT, Sheng WH, Fang CT, Hung CC, Hsieh SM, Su CP, Chiang WC, Yang JY, Lin JH, Hsieh SC, Hu HP, Chiang YP, Wang JT, Yang PC, Chang SC; SARS Research Group of the National Taiwan University/National Taiwan University Hospital. Detection of SARS-associated coronavirus in throat wash and saliva in early diagnosis. Emerg Infect Dis. 2004 Jul;10(7):1213-9. doi: 10.3201/eid1007.031113. PMID 15324540
- [Background] Watamoto T, Egusa H, Sawase T, Yatani H. Clinical evaluation of chlorine dioxide for disinfection of dental instruments. Int J Prosthodont. 2013 Nov-Dec;26(6):541-4. doi: 10.11607/ijp.3465. PMID 24179967
- [Background] Wirthlin MR, Choi JH, Kye SB. Use of chlorine dioxide mouthrinse as the ultrasonic scaling lavage reduces the viable bacteria in the generated aerosols. J West Soc Periodontol Periodontal Abstr. 2006;54(2):35-44. No abstract available. PMID 17214015
- [Background] Chen C, Zhang XJ, Wang Y, Zhu LX, Liu J. Waste water disinfection during SARS epidemic for microbiological and toxicological control. Biomed Environ Sci. 2006 Jun;19(3):173-8. PMID 16944772
- [Background] Peng X, Xu X, Li Y, Cheng L, Zhou X, Ren B. Transmission routes of 2019-nCoV and controls in dental practice. Int J Oral Sci. 2020 Mar 3;12(1):9. doi: 10.1038/s41368-020-0075-9. PMID 32127517
- [Background] Meister TL, Bruggemann Y, Todt D, Conzelmann C, Muller JA, Gross R, Munch J, Krawczyk A, Steinmann J, Steinmann J, Pfaender S, Steinmann E. Virucidal Efficacy of Different Oral Rinses Against Severe Acute Respiratory Syndrome Coronavirus 2. J Infect Dis. 2020 Sep 14;222(8):1289-1292. doi: 10.1093/infdis/jiaa471. PMID 32726430
- [Background] Shewale JG, Ratcliff JL. Overinterpretation of the antiviral results for human coronavirus strain 229E (HCoV-229E) relative to severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2). J Med Virol. 2021 Apr;93(4):1900-1902. doi: 10.1002/jmv.26722. Epub 2021 Jan 5. No abstract available. PMID 33368396

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the initial recruitment phase, 54 participants signed the consent form and were assigned to one of five study groups. However, only 49 participants completed the entire 4-week study period.
Period: Overall Study
Arm/Group | Control (Distilled Water) | Oral-B Mouth Sore (H2O2) Mouthwash | Crest Pro-Health Multi-Protection (C21H38ClN) Mouthwash | CloSYS (ClO2) Mouthwash | Listerine Mouthwash
Started | 12 | 11 | 12 | 12 | 7
Completed | 12 | 8 | 11 | 12 | 6
Not Completed | 0 | 3 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (Distilled Water) | Oral-B Mouth Sore (H2O2) Mouthwash | Crest Pro-Health Multi-Protection (C21H38ClN) Mouthwash | CloSYS (ClO2) Mouthwash | Listerine Mouthwash | Total
Number analyzed (Participants) | 12 | 11 | 12 | 12 | 7 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 11 | 10 | 11 | 9 | 7 | 48
  >=65 years | 1 | 0 | 1 | 3 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: Year] | 38.0 (11.48) | 31.7 (8.65) | 45.6 (11.77) | 45.3 (17.30) | 37.3 (12.54) | 39.9 (13.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 5 | 6 | 4 | 31
  Male | 4 | 3 | 7 | 6 | 3 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 2 | 3 | 3 | 12
  Not Hispanic or Latino | 11 | 7 | 10 | 9 | 4 | 41
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 1 | 2 | 2 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 2 | 1 | 0 | 0 | 3
  White | 7 | 4 | 6 | 6 | 5 | 28
  More than one race | 1 | 0 | 0 | 3 | 0 | 4
  Unknown or Not Reported | 0 | 4 | 2 | 1 | 2 | 9
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 12 | 12 | 7 | 54

OUTCOME MEASURES:

1. Primary Outcome: Change in SARS-CoV-2 Viral Load
Description: The change in the outcome measure, SARS-CoV-2 viral load, in saliva wash RT-PCR was measured by Cycle Threshold (Ct) value. Ct value refers to the number of cycles it takes for the fluorescent signal generated during the PCR reaction to cross a certain threshold, indicating the presence of the target nucleic acid sequence, here, SARS-CoV-2. The lower the Ct value, the faster the threshold is crossed and the higher the viral load in a biological sample, suggesting a higher concentration of the SARS-CoV-2 virus in that sample.
Time Frame: Baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: Absolute Change in Cycle Threshold
Arm/Group | Control (Distilled Water) | Oral-B Mouth Sore (H2O2) Mouthwash | Crest Pro-Health Multi-Protection (C21H38ClN) Mouthwash | CloSYS (ClO2) Mouthwash | Listerine Mouthwash
Number analyzed (Participants) | 12 | 8 | 11 | 12 | 6
Absolute Change in Cycle Threshold | -0.6 (1.9) | -0.4 (1.5) | 0.8 (1.4) | -0.4 (2.0) | -1.4 (0.8)

2. Secondary Outcome: Self-reported Clinical Symptom(s)
Description: Any self-reported (questionnaire) clinical symptom(s). A symptom checklist included cough, runny nose, scratchy/sore throat, fever, chills, fatigue, muscle ache, shortness of breath, diarrhea/nausea/vomiting, loss of taste/smell, and red /painful eye. (Clinical symptoms were collected at baseline and at 3 months; only problems with the study mouth rinse were collected daily through 4 weeks.)
Time Frame: Baseline to 3 months
Population: The denominator is the number of participants who responded to the 3 month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Control (Distilled Water) | Oral-B Mouth Sore (H2O2) Mouthwash | Crest Pro-Health Multi-Protection (C21H38ClN) Mouthwash | CloSYS (ClO2) Mouthwash | Listerine Mouthwash
Number analyzed (Participants) | 6 | 6 | 3 | 9 | 3
Participants | 1 | 0 | 0 | 0 | 0

3. Secondary Outcome: Any Hospitalization(s)
Description: Any hospitalization(s) from baseline to 4 weeks. Hospitalization(s) were collected on adverse event, unanticipated problem, and final disposition forms.
Time Frame: Baseline to 4 weeks
Population: The denominator is the number of participants who reported adverse events, unanticipated problems, or were not lost-to-follow-up before Week 4 as per final study disposition form.
Measure: Count of Participants; unit: Participants
Arm/Group | Control (Distilled Water) | Oral-B Mouth Sore (H2O2) Mouthwash | Crest Pro-Health Multi-Protection (C21H38ClN) Mouthwash | CloSYS (ClO2) Mouthwash | Listerine Mouthwash
Number analyzed (Participants) | 12 | 8 | 11 | 12 | 6
Participants | 0 | 0 | 0 | 0 | 0

4. Other Pre Specified Outcome: Change in SARS-Cov-2 Viral Load in Tobacco Users, Marijuana Smokers, or Vapers
Description: Change in saliva wash RT-PCR SARS-Cov-2 viral load in tobacco users, marijuana smokers, or vapers
Time Frame: Baseline to 4 weeks
Population: This study stopped enrollment early. The funder decided not to continue funding causing enrollment to cease and curtailing originally planned analyses. Participants with any samples collected after the baseline pre-rinse samples were included in the analysis population.
Arm/Group | Control (Distilled Water) | Oral-B Mouth Sore (H2O2) Mouthwash | Crest Pro-Health Multi-Protection (C21H38ClN) Mouthwash | CloSYS (ClO2) Mouthwash | Listerine Mouthwash
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Other Pre Specified Outcome: Change in Self-reported Clinical Symptom Onset in Tobacco Users, Marijuana Smokers, or Vapers
Description: Change in self-reported (questionnaire) clinical symptom onset in tobacco users, marijuana smokers, or vapers. A symptom checklist will include: cough, runny nose, scratchy/sore throat, fever, chills, fatigue, muscle ache, shortness of breath, diarrhea/nausea/vomiting, loss of taste/smell, and red /painful eye.
Time Frame: Baseline to 3 months
Population: as for outcome 4
Arm/Group | Control (Distilled Water) | Oral-B Mouth Sore (H2O2) Mouthwash | Crest Pro-Health Multi-Protection (C21H38ClN) Mouthwash | CloSYS (ClO2) Mouthwash | Listerine Mouthwash
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Other Pre Specified Outcome: Any Hospitalization(s) in Tobacco Users, Marijuana Smokers, or Vapers
Description: Any hospitalization(s) in tobacco users, marijuana smokers, or vapers during the study period
Time Frame: Baseline to 4 weeks
Population: as for outcome 4
Arm/Group | Control (Distilled Water) | Oral-B Mouth Sore (H2O2) Mouthwash | Crest Pro-Health Multi-Protection (C21H38ClN) Mouthwash | CloSYS (ClO2) Mouthwash | Listerine Mouthwash
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline up to 12 months.
Description: All-Cause Mortality or Serious Adverse Event
Arm/Group | Control (Distilled Water) | Oral-B Mouth Sore (H2O2) Mouthwash | Crest Pro-Health Multi-Protection (C21H38ClN) Mouthwash | CloSYS (ClO2) Mouthwash | Listerine Mouthwash
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/12 | 0/12 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/12 | 0/12 | 0/7
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/12 | 0/12 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (Distilled Water) (N=12) | Oral-B Mouth Sore (H2O2) Mouthwash (N=11) | Crest Pro-Health Multi-Protection (C21H38ClN) Mouthwash (N=12) | CloSYS (ClO2) Mouthwash (N=12) | Listerine Mouthwash (N=7)
unanticipated event (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — During sample collection on day 1, one participant used Reagent B in the DNA/RNA Shield box of ZymoResearch Company instead of distilled water in the study package for preparing the throat wash despite clear instructions with photo of steps.

LIMITATIONS AND CAVEATS:
Study support was withdrawn by Funder, so enrollment ended, and only a priori planned interim analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT04409873/Prot_SAP_000.pdf